CLINICAL TRIAL: NCT02182154
Title: Metabolism and Pharmacokinetics of [14C]-BIBF 1120 After Administration of Single Doses of 100 mg [14C]-BIBF 1120 Oral Solution in Healthy Male Volunteers
Brief Title: Metabolism and Pharmacokinetics of [14C]-BIBF 1120 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1199.20
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Healthy

ARMS (1):
- BIBF 1120 ES (Experimental)
  Interventions: Drug: BIBF 1120 ES

INTERVENTIONS:
Drug: BIBF 1120 ES

SUMMARY:
To assess the metabolic profile,

to obtain the mass balance after oral administration,

to determine the concentration of [14C]-radioactivity in blood cells, plasma, urine and faeces,

to determine BIBF 1120 and BIBF 1202 concentrations in plasma, urine, and faeces, if feasible,

to determine the protein binding of [14C]-radioactivity,

to determine the pharmacokinetics of BIBF 1120, BIBF 1202 and total radioactivity after a single oral administration of [14C]-BIBF 1120 in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects as determined by results of screening
2. Signed written informed consent in accordance with GCP and local legislation
3. Age ≥21 and ≤55 years
4. Body Mass Index ≥18.5 kg/m2 and ≤29.9 kg/m2

Exclusion Criteria:

1. Any finding of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
2. History or current gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic, hormonal disorders
3. History of any major surgery within the last four weeks before participation in this study or any bone fracture within the last two months
4. History of orthostatic hypotension, fainting spells and blackouts
5. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders
6. Chronic or relevant acute infections
7. History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
8. History of any bleeding disorder including prolonged or habitual bleeding, other haematologic disease or cerebral bleeding (e.g. after a car accident) or commotio cerebri
9. Intake of drugs with a long half-life (> 24 hours) within 1 month prior to administration
10. Planned use of any drugs which might influence the results of the trial within 10 days prior to administration or during the trial
11. Participation in another trial with an investigational drug within 2 months prior to administration or during trial
12. Smoker (> 10 cigarettes or 3 cigars or 3 pipes/day) or inability to refrain from smoking on study days
13. Alcohol abuse (> 60 g/day)
14. Drug abuse
15. Blood donation within 1 month prior to administration or during the trial
16. Excessive physical activities within 5 days prior to administration or during the trial
17. Any laboratory value outside the reference range, unless considered to lack clinical reference
18. Female gender
19. Male subjects must agree to minimize the risk of female partners becoming pregnant from the dosing day until 3 months after the completion of the study. Acceptable methods of contraception for male volunteers include a vasectomy no less than 3 months prior to dosing, barrier contraception or a medically accepted contraceptive method. For female partners of male volunteers, acceptable methods of contraception include intra-uterine device, tubal ligation, hormonal contraceptive since at least two months and diaphragm with spermicide

Ages: 21 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2005-10; Primary Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
[14C]-radioactivity in plasma and whole blood (C Blood cells/C plasma ratio of [14C]-radioactivity) | Up to 96 h after drug administration
[14C]-radioactivity in urine | Up to 120 h after drug administration
Measurement of the plasma protein binding of total [14C]-radioactivity in human plasma samples ex vivo | Up to 96 h after drug administration
Maximum observed concentration of the analyte in plasma (Cmax) | Up to 96 h after drug administration
Plasma concentration-time profiles of total radioactivity in whole blood and plasma | Up to 96 h after drug administration
[14C]-metabolic profile and identification of metabolites in urine, in comparison with various animal species | Up to 120 h after drug aministration
[14C]-radioactivity in faeces | up to 120 h after administration
[14C]-metabolic profile and identification of metabolites in faeces, in comparison with various animal species | Up to 120 h after drug aministration
[14C]-metabolic profile and identification of metabolites in plasma, in comparison with various animal species | Up to 96 h after drug aministration
Time from dosing to peak concentration (tmax) | Up to 96 h after drug administration
Terminal half-life of the analyte in plasma (t1/2) | Up to 96 h after drug administration
Terminal rate constant of the analyte in plasma (λz) | Up to 96 h after drug administration
Area under the concentration-time curve of the analyte in plasma from zero time to 24 hours (AUC0-24) | Up to 24 h after drug administration
Area under the concentration-time curve of the analyte in plasma from zero time to the time of the last quantifiable drug concentration (AUC0-tz) | Up to 96 h after drug administration
Area under the concentration-time curve of the analyte in plasma from zero time to infinity (AUC0-∞) | Up to 96 h after drug administration
Mean residence time of the analyte molecules in the body after oral administration (MRTpo) | Up to 96 h after drug administration
Total clearance of the analyte in plasma following extravascular administration (CL/F) | Up to 96 h after drug administration
Apparent volume of distribution during the terminal phase λz following extravascular administration (Vz/F) | Up to 96 h after drug administration
Fraction of analyte eliminated in urine from 0 to the limit of the last quantifiable data point (fe0-tz) | Up to 96 h after drug administration
Fraction of analyte eliminated in faeces from 0 to the limit of the last quantifiable data point (fe faeces,0-tz) | Up to 96 h after drug administration
Amount of analyte that was eliminated in faeces from 0 to the limit of the last quantifiable data point (Ae faeces,0-tz) | Up to 96 h after drug administration
Amount of analyte that was eliminated in urine from 0 to the limit of the last quantifiable data point (Ae0-tz) | Up to 96 h after drug administration

SECONDARY OUTCOMES:
Change from baseline in vital signs | Baseline, day 14 after drug administration
Change from baseline in routine laboratory | Baseline, day 14 after drug aministration
Number of participants with adverse events | Up to day 14 after drug aministration
Change from baseline in electrocardiogram | Baseline, day 14 after drug aministration
Assessment of tolerability by investigator according a 4 point scale | Day 14 after drug administration